CLINICAL TRIAL: NCT04310202
Title: A Prospective Multi-Centre Study on the Performance of the Ponto BHX Implant System
Brief Title: Multi-Centre Study on the Performance of the Ponto BHX Implant System (in Adult Patients)
Status: Completed | Type: Observational
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: Doc-00066211
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single-arm: In this single-arm study, the only interventions compared to routine clinical practice are the completion of two patient questionnaires (APHAB and GBI) and additional follow-up visits after surgery.
  Interventions: Other: Abbreviated Profile of Hearing Aid Benefit (APHAB); Other: Glasgow Benefit Inventory (GBI); Other: Additional follow-up visits after surgery

INTERVENTIONS:
Other: Abbreviated Profile of Hearing Aid Benefit (APHAB) — An intervention in this study which is outside the routine clinical practice of the clinics is the APHAB questionnaire that will be completed by the subjects on two occasions.
Other: Glasgow Benefit Inventory (GBI) — An intervention in this study which is outside the routine clinical practice of the clinics is the GBI questionnaire that will be completed by the subjects on two occasions.
Other: Additional follow-up visits after surgery — There are 1-2 additional follow-up visits after surgery (compared to the routine clinical practice of the surgeons/clinics).

SUMMARY:
This multi-centre study funded by Oticon Medical AB will be conducted at seven hospitals across Europe (UK, Spain, Denmark). Patients with a hearing loss and that are already planned for treatment with a percutaneous (through the skin) bone-anchored hearing system (BAHS) will be included in the study. A total of 50 patients will be included in the study.

The purpose of this study is to investigate the rate of successful BAHS use after implantation of the Ponto Biohelix (BHX) Implant system.

DETAILED DESCRIPTION:
This multi-centre study funded by Oticon Medical AB will be conducted at seven hospitals across Europe (UK, Spain, Denmark). Patients with a hearing loss and that are already planned for treatment with a percutaneous (through the skin) bone-anchored hearing system (BAHS) will be included in the study. A total of 50 patients will be included in the study.

The purpose of this study is to investigate the rate of successful BAHS use after implantation of the Ponto BHX Implant system. The implant, coupled to a skin-penetrating abutment, is implanted in the bone behind the ear and is later loaded with a sound processor which transforms sound waves to sound vibrations that can be sent directly to the inner ear via the skull bone. The primary objective of this study is to investigate the proportion of implant/abutment complexes providing a reliable anchorage for a sound processor, 3 months after implantation/surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients indicated for surgical intervention with a bone anchored hearing system according to local clinic's standard guidelines
* Adequate bone quality to allow for a Ponto BHX implant insertion, as judged by the investigator, and an expected bone thickness above 3 mm, where no complications during surgery are expected

Exclusion Criteria:

* Patients undergoing re-implantation
* Patients who are unable or unwilling to follow investigational procedures/requirements, e.g. to complete quality of life scales.
* Diseases or treatments known to compromise the bone quality at the implant site, e.g. radiotherapy, osteoporosis, diabetes mellitus
* Known conditions (e.g. uncontrolled diabetes) that could jeopardize skin condition and wound healing over time as judged by the investigator
* Any other known condition that the investigator determines could interfere with compliance or study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to participating clinics who meet clinical indications for surgical intervention with a bone anchored hearing system
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-17 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Implant/abutment complex capability to provide a reliable Anchorage for a sound processor | 3 months after implant surgery
  The variables assessed to determine reliable anchorage in the study are implant survival and stability, skin reactions, skin over-growth and pain preventing use of the sound processor. For a positive outcome of the primary endpoint (reliable anchorage), the implant should be in place and stable. without any adverse skin reactions or skin over-growth and pain preventing usage of the sound processor.

SECONDARY OUTCOMES:
Implant/abutment complex capability to provide reliable anchorage for sound processor | 12 months after implant surgery
  The variables assessed to determine reliable anchorage in the study are implant survival and stability, skin reactions, skin over-growth and pain preventing use of the sound processor. For a positive outcome of the primary endpoint (reliable anchorage), the implant should be in place and stable without any adverse skin reactions or skin over-growth and pain preventing usage of the sound processor.
Implant survival | 12 months after implant surgery
  Implant survival will be assessed by the investigator by means of a Yes/No question: Implant/abutment complex in place [Yes/No]
Implant stability | 12 months after implant surgery
  Clinical assessment of implant stability by the investigator by means of a Yes/No question: Implant stable [Yes/No]
Holgers score ratings | 12 months after implant surgery
  Distribution of Holgers score ratings (scale 0-4) where a higher score corresponds to a poorer outcome, assigned by investigator
IPS (Inflammation, Pain, Skin height) scores | 12 months after implant surgery
  Distribution of IPS (Inflammation [total score 0-4], Pain [score 0-2], Skin height [score 0-2]) scores assigned by investigator. The IPS score is presented as [Ix Px Sx] with x being the individual score for each parameter. A higher score corresponds to a poorer outcome
Patient-perceived presence of pain around implant/abutment | 12 months after implant surgery
  Assessment of presence of patient-perceived pain by means of a Yes/No question to the subject
Patient-perceived magnitude of pain around implant/abutment | 12 months after implant surgery
  Assessment of magnitude of patient-perceived pain using a numerical rating scale (NRS) (range 0-10) where a higher rating corresponds to a poorer outcome
Patient-perceived presence of numbness around implant/abutment | 12 months after implant surgery
  Assessment of presence of patient-perceived numbness by means of a Yes/No question to the subject
Patient-perceived magnitude of numbness around implant/abutment | 12 months after implant surgery
  Assessment of magnitude of patient-perceived numbness using a numerical rating scale (NRS) (range 0-10) where a higher rating corresponds to a poorer outcome
Skin/soft tissue overgrowth | 12 months after implant surgery
  Skin overgrowth over implant/abutment complex judged by the investigator by means of a Yes/No question
Duration of surgery | At implant surgery
  Length of surgery measured in minutes
Wound dehiscence | 12 months after implant surgery
  Prevalence of wound dehiscence measured as millimeters of dehiscence
Wound healing time | 12 months after implant surgery
  Average healing time [days] from surgery when the wound is considered healed
Implant/abutment usage | 12 months after implant surgery
  Mean hours of use of a sound processor on the implant/abutment
Subjective benefit after implant surgery | At screening visit (visit before surgery)
  Abbreviated Profile Hearing Aid Benefit (APHAB) questionnaire score (1-99) where a global higher score corresponds to a poorer outcome
Subjective benefit after implant surgery | 6 months after implant surgery
  Abbreviated Profile Hearing Aid Benefit (APHAB) questionnaire score (1-99) where a global higher score corresponds to a poorer outcome
Subjective benefit after implant surgery | 3 months after implant surgery
  Glasgow Benefit Inventory (GBI) questionnaire score (-100 to +100) where [-100] means maximum adverse effect, [0] means no effect, and [+100] means maximum positive effect
Subjective benefit after implant surgery | 12 months after implant surgery
  Glasgow Benefit Inventory (GBI) questionnaire score (-100 to +100) where [-100] means maximum adverse effect, [0] means no effect, and [+100] means maximum positive effect

OTHER OUTCOMES:
Safety outcome | 12 months after surgery
  Occurrence and severity of adverse events related to the investigational device and corresponding procedures

CONTACTS AND LOCATIONS:
Overall Officials: Rupan Banga, MD, PhD, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (6):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
- Spain (2):
  - Hospital Universitario de Donostia, San Sebastián, Gipuzkoa
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Guy's and St Thomas' NHS Foundation Trust, London